CLINICAL TRIAL: NCT04311021
Title: Current State of Impaired Awareness of Hypoglycaemia in People With Type 1 Diabetes; Change in Prevalence, Impact of Glucose Monitoring Technology and Psychosocial Impact
Brief Title: Current State of Impaired Awareness of Hypoglycaemia in People With Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: HypoResolve (Unknown)
Responsible Party: Sponsor
Other Study IDs: NL-number: NL71207.091.19
Record Dates: First submitted 2020-02-28; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-02

CONDITIONS: Diabetes type1
Keywords: Hypoglycemia; Impaired awareness of hypoglycemia; Psychosocial impact; Epidemiology
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetes type 1
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Rationale:

Hypoglycaemia is the most frequent complication of insulin treatment in individuals with type 1 diabetes and a limiting factor for achieving optimal glycaemic control. When recurrent, hypoglycaemia can induce a process of habituation, leading to impaired awareness of hypoglycaemia (IAH), a process that can be reversed by meticulous avoidance of hypoglycaemia. In the past 5-10 years, the use of continuous real-time (RT-CGM) or flash glucose monitoring (FGM) has increased rapidly in the clinical management of type 1 diabetes to improve overall glycaemic control and reduce the frequency of hypoglycaemic events, in particular in patients with IAH. It is unknown, however, whether the use of these devices, as well as other improvements in clinical management, has reduced the prevalence IAH and exposure to severe hypoglycaemia (SH) in subjects with type 1 diabetes in a real-world setting. Therefore, it becomes highly appropriate to investigate the current state of IAH and SH in type 1 diabetes. Also, since invites to this study will specifically include people who have taken part of previous assessments, this study will be able to investigate the change in IAH over time and the potential contributing role of RT-CGM/FGM. Furthermore, we want to explore associations of IAH and SH with clinical parameters, quality of life and psychosocial impact. This knowledge will help people with diabetes and their healthcare providers to better adjust treatment recommendations to individual targets.

Objective:

The primary objective of our study is to investigate the current prevalence of IAH and exposure to severe hypoglycaemia in individuals with diabetes type 1.

The secondary objectives of our study are to:

* Study the difference in IAH prevalence over time in individuals with diabetes type 1.
* Assess the association of RT-CGM/FGM with IAH and SH.
* Study thoughts, emotions and worries which lead to a certain behaviour in case of hypoglycaemia and prevention of hypoglycaemia.
* Study associations of IAH and history of SH with productivity in different situations (work/study, relation/sexuality, driving behaviour/traffic and sport/leisure).
* Study association between partner involvement and handling in case of (unawareness for) hypoglycaemia.
* Study knowledge of subjects with diabetes about hypoglycaemia and IAH.
* Study burden of IAH and severe hypoglycaemia on family members of people with type 1 diabetes, as experienced by patients themselves.

Study design:

This study will be a cross-sectional observational cohort study. The study will be conducted at the Radboud university medical center, department of internal medicine. Subjects with type 1 diabetes will be recruited from outpatient diabetes clinic as well as subjects who participated in two earlier cohorts and agreed to be approached again.

Study population:

The study population will be individuals with diabetes type 1, older than sixteen years old.

Main study parameters/endpoints The main study parameter will be the current prevalence of IAH and exposure to severe hypoglycaemia in the past 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes diagnosis based on clinical judgement with or without auto-antibodies, according to the ISPAD Clinical Practice Consensus Guidelines 2018 (27). Briefly, clinical criteria for the diagnosis of diabetes mellitus include an acute presentation, classical symptoms of diabetes or profound hyperglycaemia with or without ketoacidosis, a plasma glucose concentration ≥11.1 mmol/L and considerably elevated HbA1c, and age of onset >6 months.
* Age ≥16 years.
* Ability to provide written informed consent.
* Fluency in speaking and reading Dutch.

Exclusion Criteria:

* Severe psychiatric comorbidity that leads to inability to provide informed consent or as judged by the healthcare provider
* Other comorbidity interfering with completing surveys, as judged by the healthcare professional.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with diabetes type 1.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-01-23 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
The main study parameter will be the current prevalence of IAH and exposure to SH in the past 12 months. | Past 12 months

SECONDARY OUTCOMES:
Difference in IAH prevalence over the years. | Past 12 years.
Relationship between IAH/SH prevalence and RT-CGM/FGM vs traditional glucometer use. | Past 12 months.
Answers to questionnaire | Past 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://hypo-resolve.eu/